CLINICAL TRIAL: NCT02003586
Title: Effect of a Plant-based Ingredient on Generalized Hormonal Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FDS-NAA-1462
Record Dates: First submitted 2013-11-22; First posted 2013-12-06 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: subjects

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plant-based ingredient to a starchy meal (Other): Plant-based ingredient
  Interventions: Dietary Supplement: plant-based ingredient; Dietary Supplement: No plant-based ingredient
- Starchy meal alone (Other): No plant-based ingredient
  Interventions: Dietary Supplement: plant-based ingredient; Dietary Supplement: No plant-based ingredient

INTERVENTIONS:
Dietary Supplement: plant-based ingredient
Dietary Supplement: No plant-based ingredient

SUMMARY:
The study is designed to determine the extent to which foods containing a plant-based ingredient affect blood glucose and hormonal response in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, Age at start of the study >20 and <50 years;
* Body mass index (BMI) ≥ 20,0 and ≤ 25,0 kg/m2;
* Apparently healthy: no medical conditions which might affect the study measurements, absorption, metabolism and distribution (including diabetes type 1 and type 2, gastrointestinal dysfunction, gastrointestinal surgery and inflammatory diseases);
* Fasting blood glucose value of subjects is ≥ 3.4 and ≤ 6.1 mmol/litre (i.e. 62-110 mg/dl) at screening;
* Agreeing to be informed about medically relevant personal test-results by a physician;
* Informed consent signed;
* Willing to comply to study protocol during study;
* Covered by Health Insurance System and/or in compliance with the recommendations of National Law in force relating to biomedical research.
* Accessible veins on arms as determined by examination at screening.

Exclusion Criteria:

* Any history of diabetes, hyper- (or hypo-) glycemia or other disorder of glucose metabolism;
* Blood donation in the past 2 months;
* Reported participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study;
* Reported participation in night shift work two weeks prior to pre-study investigation or during the study. Night work is defined as working between midnight and 6.00 AM;
* Reported intense sporting activities > 10h/w;
* Consumption of > 21 alcoholic drinks in a typical week;
* Not being used to eat breakfast;
* Reported use of any nicotine containing products in the six months preceding the study and during the study itself;
* Use of medication which interferes with study measurements;
* Reported dietary habits: medically prescribed diet, slimming diet;
* Not used to eat 3 meals a day;
* Vegetarian;
* Reported weight loss/gain (>10%) in the last six month before the study;
* Being an employee of Unilever and CRO;
* Allergy or intolerance to food products and aversion to food products provided during the study;
* Subject who cannot be contacted in case of emergency;
* Subject who, in the judgment of the investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
* Subject under guardianship;
* Subject who would receive more than 4500 euro's as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
AUC of post-prandial hormones | 120 minutes
  Amylin (total) will be assessed.
AUC of post-prandial hormones | 120 minutes
  Ghrelin (active) will be assessed.
AUC of post-prandial hormones | 120 minutes
  Glucose-dependent insulinotropic peptide (gastric inhibitory polypeptide, GIP) (total) will be assessed.
AUC of post-prandial hormones | 120 minutes
  Glucagon-like peptide-1 (GLP-1) (active) will be assessed.
AUC of post-prandial hormones | 120 minutes
  Leptin will be assessed.
AUC of post-prandial hormones | 120 minutes
  Pancreatic polypeptide (PP) will be assessed.
AUC of post-prandial hormones | 120 minutes
  Peptide YY (PYY) (total) will be assessed.
AUC of post-prandial hormones | 120 minutes
  Insulin will be assessed.
AUC of post-prandial hormones | 120 minutes
  C-peptide will be assessed.
AUC of post-prandial hormones | 120 minutes
  Glucagon will be assessed.

SECONDARY OUTCOMES:
AUC of post-prandial hormones | 180 and 240 minutes
  Amylin (total) will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  Ghrelin (active) will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  Glucose-dependent insulinotropic peptide (gastric inhibitory polypeptide, GIP) (total) will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  Pancreatic polypeptide (PP) will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  Peptide YY (PYY) (total) will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  Leptin will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  Glucagon will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  Insulin will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  C-peptide will be assessed.
AUC of post-prandial hormones | 180 and 240 minutes
  Glucagon-like peptide-1 (GLP-1) (active) will be assessed.

OTHER OUTCOMES:
Blood glucose response (+iAUC) | 120 and 180 minutes
  Effect on blood glucose response.

CONTACTS AND LOCATIONS:
Overall Officials: Yves DONAZZOLO, M.D., M.Sc., Principal Investigator — EUROFINS OPTIMED, GIERES - France
Locations (1):
- Eurofins Optimed Clinical research, Gières, France